CLINICAL TRIAL: NCT01360697
Title: A Multi-Centre Demonstration Project to Evaluate the Effectiveness and Acceptability of the Joint Asia Diabetes Evaluation (JADE) in Chinese Type 2 Diabetic Patients in Jiangsu and Anhui (JA), China
Brief Title: An Evaluation of the Effectiveness and Acceptability of Delivering Structured Care in Chinese Type 2 Diabetic Patients
Acronym: JADE-JA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asia Diabetes Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2011-095-T
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes
Keywords: Diabetes; Structured care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- JADE- JA (Experimental): Use the JADE portal to monitor the delivery of structured care.
  Interventions: Other: JADE
- Usual care (Active Comparator): Patients will receive usual care in between two annual comprehensive assessments.
  Interventions: Other: Non-JADE

INTERVENTIONS:
Other: JADE — 1. The nurse will complete the CA using standardized protocol including blood & urine tests, eye & feet examination.
  2. Whenever feasible, the nurse will arrange 2-4 hours of diabetes education in groups or on an individual basis as appropriate.
  3. Between each follow-up (FU) visit, the nurse or HCA will contact the patient by phone or email to remind them to attend visits, adhere to medications & healthy lifestyles, perform self blood glucose monitoring as appropriate.
  4. At each FU visit, the patients will first see the nurse or HCA for record of blood pressure, body weight & blood glucose (or A1c) measurement as appropriate. Compliance will also be checked using the 4-item questionnaire.
  5. After the FU visit, the patients will see the nurse or HCA again to clarify any issues & concerns, reinforce compliance & record any changes in medications.
  6. After each FU visit, the HCA will generate summary reports to be given to patients & doctors to promote sharing of information.
  Arms: JADE- JA
Other: Non-JADE — Patients will receive a comprehensive assessments at baseline and again after 12 months. In the interim between these two time points patients will be managed according to 'usual care' procedures.
  Arms: Usual care

SUMMARY:
In this demonstration project (JADE in Jiangsu & Anhui Program, JADE-JA in short) led by key opinion leaders in the field of diabetes and endocrinology in Jiangsu and Anhui area and supported by the ADF, shall recruit 4800 type 2 diabetic patients attending medical out-patient clinics in the area to compare the effects of usual versus structured care (non-JADE vs JADE) on metabolic control, quality of life and behavioral changes. After explanation by trained doctors and nurses and with written informed consent, patients will be randomized to either the JADE or non-JADE group. The former encompasses all components of the structured care delivered by a trio-team of doctor, nurse and Healthcare Assistant (HCA) while the non-JADE group only consists of comprehensive assessments (CA) at baseline and 12-month with patients managed in the usual manner thereafter. At the end of 12 months, all patients will undergo repeat comprehensive assessments for comparison of rates of attainment of treatment targets, behavioral changes, quality of life and default rates. The acceptability of the JADE-JA Program by patients and the trio-team will also be evaluated.

The investigators hypothesize that the use of state of the art information technology to record, manage and analyze the large amount of clinical information generated during various consultation visits will improve the effectiveness and efficiency in implementing these care protocols through decision support and regular feedback to both patients and care team.

DETAILED DESCRIPTION:
In 2007, supported by an educational grant, a charitable organization named the Asia Diabetes Foundation (ADF) (www.adf.org.hk) was established to develop the Joint Asia Diabetes Evaluation (JADE) Program, which comprises a web-based disease management program to enable doctors, nurses and other care personnel to manage people with diabetes in an integrated and effective manner. The JADE electronic portal (e portal) provides a virtual platform to facilitate implementation of evidence-based clinical protocols with ongoing data collection, management and analysis to track performance for quality assurance and improvement purposes. The JADE Program also incorporates validated risk equations developed by the Chinese University of Hong Kong (CUHK) Diabetes Care & Research Group to stratify patients into various risk levels for recommendation of triage into different care protocols with decision supports. This clinical information, presented in the forms of charts and time trends, can be communicated to patients and care providers to motivate behavioral changes, set treatment goals and attain targets.

By participating in the JADE Program, the doctors will be able to create their own diabetes registry to benchmark their performance including adherence to procedures, recall of default patients and rate of attainment of treatment targets. In this regard, the implementation of the full JADE Program requires changes in the practice environment and deployment of additional manpower (e.g. a nurse and a HCA) to enter data and provide reminders to patients and doctors to improve adherence to protocols.

It is anticipated that the cost-effectiveness of the structured (JADE group) versus usual (non-JADE group) care on rates of attainment of multiple treatment targets, which will translate into clinical outcomes in the long term, will eventually change practice and policy to make quality diabetes care more affordable, sustainable and accessible in China.

In this 1-year multi-centre randomized study, the investigators shall use a web-based disease management program (JADE e portal) to facilitate implementation of structured care with the following objectives:

* To evaluate the reach, adoption and acceptability of the JADE e portal by patients and health care team
* To compare the effectiveness of the JADE versus non-JADE Program in attainment of treatment targets, improvement of quality of life and changes in behaviours
* To document the pattern of complications, risk factors, use of medications and quality of life in type 2 diabetic patients in Jiangsu and Anhui, China.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients attending the 8 hospitals or affiliated clinics led by PIs of the JADE-JA Program who are living in the area with an intention to have 'regular' follow-up
* Aged ≥ 18 years
* Patients can have newly diagnosed or established disease, treated with lifestyle or blood glucose lowering drugs including oral agents with or without insulin
* For newly diagnosed type 2 diabetic patients, their plasma glucose levels should be:

  * Fasting plasma glucose (PG) ≥ 7.0 mmol/L on 2 or more occasions, and/or
  * Random (or post-OGTT 2h) PG ≥ 11.1 mmol/L on 2 or more occasions, and/or

Exclusion Criteria:

* Type 1 diabetes defined as a history of ketosis at diagnosis [acute symptoms with heavy ketonuria (> 3+) or ketoacidosis] or continuous requirement of insulin within one year of diagnosis
* Patients with reduced life expectancy (e.g. less than 6-months) due to recent diagnosis of advanced cancers (e.g. within last 2 years) and other life threatening conditions
* Patients with a mental condition rendering them unable to understand the nature, scope, and possible consequences of the study
* Patients actively enrolled in another intervention study
* Patients who are unwilling to return for regular follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who attain 2 or more of the 'ABC'targets | 12 months
  Percentage of patients who attain 2 or more of the following 3 targets:
  1. HbA1c <7%
  2. BP <130/80 mmHg
  3. LDL cholesterol <2.6 mmol/L

SECONDARY OUTCOMES:
New onset of all diabetes-related endpoints | 12 months
  This includes:
  1. cardiovascular endpoints (acute myocardial infarction, revascularisation procedures, heart failure or unstable angina or arrhythmia requiring hospital admissions, stroke, lower extremity amputation or foot ulcers);
  2. chronic kidney disease (eGFR<60 ml/min/1.73m2) and end stage renal disease (dialysis and/or eGFR<30;ml/min/1.73m2)
  3. visual impairment (corrected visual acuity of 20/200 or lower) or eye surgery;
  4. cancer
  5. any hospitalization due to complications related to diabetes and/or its treatment (such as hypoglycaemic attacks)
  6. death
Quality of Life | 12 Months
Behavioral changes (in the last 3 months) | 12 months
  1. Frequency of Self Blood Glucose Monitoring (SBGM)
  2. Adherence to balanced eating
  3. Adherence to regular exercise
  4. Adherence to recommended procedures (e.g. return for blood tests or education classes)
Frequency of hypoglycaemia (in the last 3 months) | 12 months
Number of hospitalizations, follow up visits by doctors and other care professionals during the 12 months | 12 months
Default rates at the end of the study | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Chan, MD, Principal Investigator — Asia Diabetes Foundation; Gary Ko, MD, Principal Investigator — Asia Diabetes Foundation
Locations (8):
- China (8):
  - Chinese Medicine Hospital of Anhui Province, Anhui
  - Third People's Hospital of Hefei City, Hefei
  - HuaiAn Second People's Hospital, HuaiAn
  - Jiangsu Province Official Hospital, Jiangsu
  - Rehab Hosp of Zhenjiang, Jiangsu Province, Jiangsu
  - The Affiliated Hosp of Jiangsu-Nantong U, Jiangsu
  - First People's Hospital of Kunshan City, Kunshan
  - Second Affiliated Hospital of Suzhou University, Suzhou

REFERENCES:
- See also: Works of the Asia Diabetes Foundation, including JADE-JA program — http://www.adf.org.hk